CLINICAL TRIAL: NCT04212104
Title: The Effect of Watching Mukbang on the Desire to Eat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1806008044
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Mukbang
Keywords: mukbang; randomized and controlled trail; desire to eat

STUDY DESIGN:
Intervention Model Description: The study randomly assigned participants to watch either a mukbang, or a non-food content video. Participants report their attitudes such as satiation and disgust, and report their desire to eat several kinds of foods after watching the assigned video.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- watch mukbang (Experimental): participants are assigned to watch a dim sum mukbang by a famous host, Peggie Neo (https://youtu.be/2dRf535eAPK, accessed: 2018-9-12)
  Interventions: Other: watch a mukbang
- watch non-food content video (Placebo Comparator): participants are assigned to watch the Big Bang Theory, The Euclid Alternative ( https://youtu.be/V8kUL9owk6Q, accessed: 2018-9-12).
  Interventions: Other: watch a non-food video

INTERVENTIONS:
Other: watch a mukbang — watch the dim sum mukbang
  Arms: watch mukbang
Other: watch a non-food video — watch the Big Bang Theory video
  Arms: watch non-food content video

SUMMARY:
The current study is designed to find the effect of mukbang on dieters. Mukbang is an online eating broadcast where a host (Asian mukbangs generally feature a young and slim female host) consumes a large amount of food while chatting with audiences. Since some dieters watch mukbang to get satiation and control their appetites, the investigators proposed the hypothesis that mukbang could increase people's satiation level and decrease their desire to eat. To test this hypothesis, one randomized controlled study was conducted and female participants were randomly selected to watch either a mukbang or a non-food related video. Their desire to eat were reported and measured after the video.

ELIGIBILITY:
Inclusion Criteria:

* Female, English native speakers

Exclusion Criteria:

* Male, English is not mother language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
satiation | report the feeling right after the intervention (since participants were first randomized to watch a video when participated in the study, after the intervention, i.e., after the video means 3 minutes after participants started the study)
  participants report their satiation level, on a scale from -3 to 3. -3 means not satisfied at all, 3 means very satisfied.
disgust | report the feeling right after the intervention (since participants were first randomized to watch a video when participated in the study, after the intervention, i.e., after the video means 3 minutes after participants started the study)
  participants report their disgust level, on a scale from -3 to 3. -3 means not disgust at all, 3 means very disgust
desire to eat dim sum | report the feeling right after the intervention (since participants were first randomized to watch a video when participated in the study, after the intervention, i.e., after the video means 3 minutes after participants started the study)
  participants report their desire to eat dim sum, on a scale from 0 to 10. 0 means not want to eat dim sum at all, 10 means very want to eat dim sum.
desire to eat fruits or vegetables | report the feeling right after the intervention (since participants were first randomized to watch a video when participated in the study, after the intervention, i.e., after the video means 3 minutes after participants started the study)
  participants report their desire to eat fruits or vegetables, on a scale from 0 to 10. 0 means do not want to eat fruit or vegetable at all, 10 means very want to eat fruit or vegetable.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided